CLINICAL TRIAL: NCT06059339
Title: Comparing Postoperative Opioid Consumption of Pericapsular Nerve Group (PENG) Block with Lumbar Erector Spinae Plain Block in Total Hip Arthroplasty Surgery
Brief Title: Comparing Pericapsular Nerve Group Block with Lumbar Erector Spinae Plain Block in Total Hip Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Beliz Bilgili, Associated Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 01.2023.886
Record Dates: First submitted 2023-04-04; First posted 2023-09-28 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain; Total Hip Arthroplasty
Keywords: Total Hip Arthroplasty; PENG Block; Lumbar Erector Spinae Plain Block; Postoperative Opioid Consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PENG Block and Spinal Anesthesia (Active Comparator): The patients receive PENG block with 20 ml 0,25% bupivacaine for postoperative pain management at the beginning of the surgery. Before the block performance, patients received spinal anesthesia at the L3-L4 level with 20 mg heavy bupivacaine. All patients will receive the same postoperative multimodal analgesia regimen, which includes intravenous paracetamol 1000 mg every 6 hours and intramuscular diclofenac 75 mg every 12 hours. In addition, intravenous patient-controlled analgesia (PCA) with morphine will be administered for 48 hours postoperatively, with a bolus dose of 1 mg and a lockout interval of 10 minutes (no basal rate). If the Numeric Rating Scale (NRS) exceeds 4, intravenous tramadol (1.5 mg/kg) will be administered as rescue analgesia.
  Interventions: Other: Procedure/Surgery: Regional Block Comparison Comparing postoperative pain and opioid consumption in groups
- Lumbar Erector Spinae Plain Block and Spinal Anesthesia (Active Comparator): The patients receive LESP block for postoperative pain management at the beginning of the surgery. The LESP block will be provided with 40 ml 0,25% bupivacaine under ultrasonography. Following the block performance, patients received spinal anesthesia at the L3-L4 level with 20 mg heavy bupivacaine. All patients will receive the same postoperative multimodal analgesia regimen, which includes intravenous paracetamol 1000 mg every 6 hours and intramuscular diclofenac 75 mg every 12 hours. In addition, intravenous patient-controlled analgesia (PCA) with morphine will be administered for 48 hours postoperatively, with a bolus dose of 1 mg and a lockout interval of 10 minutes (no basal rate). If the Numeric Rating Scale (NRS) exceeds 4, intravenous tramadol (1.5 mg/kg) will be administered as rescue analgesia.
  Interventions: Other: Procedure/Surgery: Regional Block Comparison Comparing postoperative pain and opioid consumption in groups
- PENG Block and Lumbar Erector Spinae Plain Block and Spinal Anesthesia (Active Comparator): The patients receive LESP block and PENG block for postoperative pain management at the beginning of the surgery. The LESP block (40 ml) and PENG block (20 ml) will be provided with 0,25% bupivacaine each under ultrasonography. Patients receive spinal anesthesia at the L3-L4 level with 20 mg heavy bupivacaine. All patients will receive the same postoperative multimodal analgesia regimen, which includes intravenous paracetamol 1000 mg every 6 hours and intramuscular diclofenac 75 mg every 12 hours. In addition, intravenous patient-controlled analgesia (PCA) with morphine will be administered for 48 hours postoperatively, with a bolus dose of 1 mg and a lockout interval of 10 minutes (no basal rate). If the Numeric Rating Scale (NRS) exceeds 4, intravenous tramadol (1.5 mg/kg) will be administered as rescue analgesia.
  Interventions: Other: Procedure/Surgery: Regional Block Comparison Comparing postoperative pain and opioid consumption in groups

INTERVENTIONS:
Other: Procedure/Surgery: Regional Block Comparison Comparing postoperative pain and opioid consumption in groups — Procedure/Surgery: Regional Block Comparison Comparing postoperative pain and opioid consumption in groups

SUMMARY:
Total hip arthroplasty is a common surgical procedure aiming to improve mobility and quality of life in patients suffering from hip pain. Despite being a frequently performed procedure, there is high variability in the peri-operative anaesthetic and analgesic management for total hip arthroplasty.

Beyond the immediate postoperative period, regional anesthesia and analgesia can have potentially beneficial effects on long-term outcomes, especially on postoperative pain, functional rehabilitation and morbidity .

The primary implication of this study is to compare postoperative opioid consumption of patients' after total hip arthroplasty using pericapsular nerve group (PENG) block with lumbar erector spinae plain block.

DETAILED DESCRIPTION:
Total hip arthroplasty is a common surgical procedure aiming to improve mobility and quality of life in patients suffering from hip pain. Despite being a frequently performed procedure, there is high variability in the peri-operative anaesthetic and analgesic management for total hip arthroplasty.

Beyond the immediate postoperative period, regional anesthesia and analgesia can have potentially beneficial effects on long-term outcomes, especially on postoperative pain, functional rehabilitation and morbidity .

The primary implication of this study is to compare postoperative opioid consumption of patients' after total hip arthroplasty using pericapsular nerve group (PENG) block with lumbar erector spinae plain block.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, undergoing total hip arthroplasty surgery

Exclusion Criteria:

* Patients with solid organ dysfunction, chronic opioid or corticosteroid use, bleeding diathesis, patients receiving inpatient medication, patients with psychiatric disorders and patients who cannot be contacted after surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-04-22 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | 24 Hours
  Comparing opioid consumption via Patient Controlled Analgesia (PCA) device
  1 mg/ ml morphine, 10 minutes lock out

SECONDARY OUTCOMES:
Pain Scores | 48 Hours
  Numeric Rating Scale: (0 to 10: worse pain:10 no pain:0)
rescue analgesia | 48 hours
  tramadol 1.5 mg/kg if NRS>4.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided